CLINICAL TRIAL: NCT02309372
Title: A Randomized, Controlled Pilot Trial Assessing the Utility of Cognitive Behavioral Therapy to Improve Endothelial Function and Reduce Inflammation in Depressed, Virologically-Suppressed, Antiretroviral-Treated, HIV-infected Adults
Brief Title: Depression Therapy to Improve Cardiovascular Risk in HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Samir K Gupta, MD, MS, Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HL126557 (NIH)
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Results first posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Depression; HIV
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Behavioral Therapy (CBT) (Experimental): Those assigned to the CBT arm will undergo therapy with the Beating the Blues (BtB) computerized intervention.
  Interventions: Behavioral: Beating the Blues
- Usual Care (No Intervention): No specific depression care will be provided through this study for those assigned to this arm. However, the participant's caregiver may choose to provide depression treatment outside of this trial.

INTERVENTIONS:
Behavioral: Beating the Blues — Computerized depression treatment intervention
  Arms: Cognitive Behavioral Therapy (CBT)

SUMMARY:
This trial will determine if depression treatment will reduce cardiovascular risk in HIV-infected patients already receiving HIV treatments. Half of the participants will undergo a specific computerized depression treatment with the other half receiving usual care from their HIV providers.

DETAILED DESCRIPTION:
The objectives of this study will be met by performing a 24-week, randomized, controlled, single-blinded, two-arm, parallel group, pilot trial at a single center. A total of 200 subjects may be screened to identify 110 participants to be enrolled and randomized. These participants will be ≥ 18 years old, have been receiving antiretroviral therapy for at least one year with an HIV viral load < 75 copies/mL at screening, and have major depression using the PHQ-9 questionnaire. These participants will be randomized 1:1 to either depression treatment with the Beating-the-Blues cognitive behavioral therapy program (N=55) or usual care (N=55).

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, documented by both: (1) any licensed rapid HIV test or HIV enzyme test kit at any time prior to study entry and (2) by at least one detectable HIV-1 antigen or at least one detectable plasma HIV-1 RNA viral load
* Age equal to or greater than 18 years
* Receipt of antiretroviral therapy of any kind for at least 360 days prior to screening

Note: Interruptions in ART of up to 14 days total during the 360 days prior to screening are allowed

* HIV-1 RNA level < 75 copies/mL at screening

NOTE: There are no CD4 cell count eligibility criteria for this trial

* For women who are still of reproductive potential, a negative urine pregnancy test
* Depression as defined by having a score ≥ 10 on the PHQ-9 questionnaire

Exclusion Criteria:

* Inability to complete written, informed consent
* Incarceration at the time of any study visit
* Active suicidality, as determined by the patient's HIV provider or social worker following a positive response (1, 2, or 3) to PHQ-9 Item #9 and a positive response (yes) to one or more of the three questions on the Patient Suicidality Form (with last suicide attempt within the past ten years)
* Diagnosed vascular disease (documented history of angina pectoris, coronary disease, peripheral vascular disease, cerebrovascular disease, aortic aneurysm, or otherwise known atherosclerotic disease)
* History of congestive heart failure, even if currently compensated
* Diagnosed disease or process, besides HIV infection, associated with increased systemic inflammation (including, but not limited to, systemic lupus erythematosis, inflammatory bowel diseases, other collagen vascular diseases)

Note: Hepatitis B or C co-infections are NOT exclusionary

* Known or suspected malignancy requiring systemic treatment within 180 days of screening

NOTE: Localized treatment for skin cancers is not exclusionary

* History of Raynaud's phenomenon
* History of cardiac arrhythmias or cardiomyopathy
* Uncontrolled hyperthyroidism or hypothyroidism, defined as TSH values outside of the local reference range on most recent clinical assessment
* History of carotid bruits
* Systolic blood pressure > 160 mmHg or diastolic blood pressure > 110 mmHg at screening
* Screening estimated glomerular filtration rate (eGFR) < 50 mL/min/1.732 (using the 2009 CKD-EPI equation) using a serum creatinine level measured at screening
* Screening glucose ≥ 140 mg/dL or hemoglobin A1c > 8.0%
* Screening total cholesterol > 240 mg/dL
* Therapy for serious medical illnesses within 14 days prior to screening

Note: Therapy for serious medical illnesses that overlaps with a main study visit will result in postponement of that study visit until the course of therapy is completed; postponement outside of the allowed study visit timeframe will result in study discontinuation

* Pregnancy or breastfeeding during the course of the study
* Receipt of investigational agents, cytotoxic chemotherapy, systemic glucocorticoids (of any dose), or anabolic steroids at screening

Note: Physiologic testosterone replacement therapy or topical steroids is not exclusionary. Inhaled/nasal steroids are not exclusionary as long as the participant is not also receiving HIV protease inhibitors

* Active drug use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements
* History of schizophrenia or bipolar disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir K Gupta, MD, Principal Investigator — Indiana University School of Medicine; Jesse C Stewart, PhD, Principal Investigator — Indiana University School of Medicine
Locations (2):
- United States (2):
  - Indiana University Health University Hospital, Indiana Clinical Research Center, Indianapolis, Indiana
  - Infectious Diseases Research Center, Indianapolis, Indiana

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognitive Behavioral Therapy (CBT) | Usual Care
Started | 27 | 27
Completed | 24 | 25
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Therapy (CBT) | Usual Care | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (9.8) | 45.6 (11.9) | 45.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 23 | 22 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 15 | 36
  White | 6 | 10 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Brachial Artery Flow-mediated Dilation From Baseline to Week 12
Description: Changes in flow-mediated dilation of the brachial artery from baseline to week 12. This is calculated by the FMD value at Week 12 minus the FMD value at baseline.
Time Frame: Baseline and Week 12 of participation
Measure: Mean (Standard Deviation); unit: absolute percent change
Arm/Group | Cognitive Behavioral Therapy (CBT) | Usual Care
Number analyzed (Participants) | 24 | 25
absolute percent change | -0.47 (2.65) | 0.29 (2.93)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy (CBT) vs Usual Care; Test type: Superiority; p = 0.32, t-test, 2 sided; Mean Difference (Net) = -0.76, 95% CI 2-sided [-2.28 to 0.77]

2. Secondary Outcome: Changes in Circulating IL-6 From Baseline to Week 12
Description: Interleukin-6 (IL-6) is a measure of systemic inflammation. This is calculated by the IL-6 value at Week 12 minus the IL-6 value at baseline.
Time Frame: Baseline and 12 weeks
Population: Participants who had blood samples available for analysis at both baseline and Week 12
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Cognitive Behavioral Therapy (CBT) | Usual Care
Number analyzed (Participants) | 23 | 24
pg/mL | 2.38 (8.71) | 1.24 (4.16)

3. Secondary Outcome: Change in hsCRP From Baseline to Week 12
Description: hsCRP (high sensitivity C-reactive protein) is a measure of systemic inflammation. This is calculated by the hsCRP value at Week 12 minus the hsCRP value at baseline.
Time Frame: 12 weeks
Population: Participants who had blood samples available for analysis at both baseline and Week 12
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Cognitive Behavioral Therapy (CBT) | Usual Care
Number analyzed (Participants) | 23 | 24
mg/L | 1.22 (3.89) | 1.06 (4.71)

4. Secondary Outcome: Change in D-dimer From Baseline to Week 12
Description: D-dimer is a measure of systemic coagulation. This is calculated by the D-dimer value at Week 12 minus the D-dimer value at baseline.
Time Frame: 12 weeks
Population: Participants who had blood samples available for analysis at both baseline and Week 12
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cognitive Behavioral Therapy (CBT) | Usual Care
Number analyzed (Participants) | 23 | 24
ng/mL | 3.69 (466) | -10.26 (651)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Cognitive Behavioral Therapy (CBT) | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 5/27 | 1/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cognitive Behavioral Therapy (CBT) (N=27) | Usual Care (N=27)
Suicidal ideation (Psychiatric disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Elevated creatine kinase (Musculoskeletal and connective tissue disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alcohol abuse (Psychiatric disorders) | 1 | 0
Arthroplasty of toe (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT02309372/Prot_SAP_000.pdf